CLINICAL TRIAL: NCT03537352
Title: Shared Decision Making in Patients With Surgical or Non-Surgical Diseases in a General Hospital: A Pilot Study
Brief Title: Shared Decision Making in a General Hospital
Status: Completed | Type: Observational
Sponsor: Psychiatric Hospital of Attica (Other)
Collaborators: Thriasio General Hospital of Elefsina (Other)
Responsible Party: Principal Investigator, Dimitrios Kontis, Department Head, 4th Psychiatric Department, Psychiatric Hospital of Attica
Other Study IDs: PsychiatricHA
Record Dates: First submitted 2018-05-15; First posted 2018-05-25 (Actual); Last update posted 2018-11-27 (Actual); Status verified 2018-11

CONDITIONS: Surgical Procedure, Unspecified; General Medical Condition

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Surgical Disorders: A. Surgical Disorders:
  1. Current Hospitalization at the Surgical Inpatient Department or at the Inpatient Department of Otorhinolaryngology or at the Inpatient Department of Cardiology OR
  2. Current Follow-up at the Surgical Outpatient Department or at the Outpatient Department of Otorhinolaryngology or at the Outpatient Department of Cardiology due to a disorder for which any appropriate surgical treatment (surgery) is a treatment option.
  Interventions: Procedure: Any appropriate surgical treatment
- Non-Surgical General Medical Disorders: 1. Current Hospitalization at the Internal Medicine Inpatient Department or at the Inpatient Department of Cardiology OR
  2. Current Follow-up at the Internal Medicine Outpatient Department or at the Outpatient Department of Cardiology due to a disorder for which surgery is not a treatment option and any appropriate drug or non-drug treatment excluding surgery is a treatment option.
  Interventions: Drug: Any appropriate drug or non-drug treatment excluding surgery

INTERVENTIONS:
Procedure: Any appropriate surgical treatment — Any appropriate surgical treatment for the management of patient's current disorder
  Groups: Surgical Disorders
Drug: Any appropriate drug or non-drug treatment excluding surgery — Any appropriate drug or non-drug treatment excluding surgery for the management of patient's current disorder
  Groups: Non-Surgical General Medical Disorders

SUMMARY:
A pilot cross-sectional study will investigate the differential effect of the type of disorder (surgical versus non-surgical) on the scores of the 9-item shared decision making questionnaire.

DETAILED DESCRIPTION:
During a pilot cross-sectional study, the 9- Item Shared Decision Making Questionnaire (9SDMQ) will be administered in two groups of participants, one (N=60) suffering from surgical diseases and one (N=60) from non-surgical medical diseases. Patients hospitalized in four acute wards (2 surgical and 2 non-surgical wards) or visiting the relevant outpatient departments of the Triassion General Hospital of Elefsina, Greece will be recruited. The primary outcome will be the difference on the 9SDMQ scores (transformed in a 1-100% scale) in patients suffering from surgical versus non-surgical disorders. Secondary outcome measures will include the effect of patients' demographic and clinical variables, of physicians' demographic variables and of the score on the Montreal Cognitive Assessment on the 9SDMQ scores. Additionally the relationship of patients' satisfaction on the 9SDMQ scores will also be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Hospitalization in the Thriassion General Hospital of Elefsina
* Ability to give informed consent

Exclusion Criteria:

* Inability to complete the neuropsychological assessment
* Mental retardation

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients hospitalized in 4 acute wards (2 for surgical and 2 for non-surgical disorders) or the relevant outpatient departments
Sampling Method: Non-Probability Sample
Enrollment: 120 (Actual)
Dates: Start 2018-05-14 (Actual); Primary Completion 2018-11-21 (Actual); Study Completion 2018-11-21 (Actual)

PRIMARY OUTCOMES:
Difference in scores of the 9-Item Shared Decision Making Questionnaire between surgical and non-surgical disorders | one year
  Difference in scores of the 9-Item Shared Decision Making Questionnaire between surgical and non-surgical disorders

SECONDARY OUTCOMES:
Effect of patients' age, education, gender, maternal education, nationality on 9-item SDM Questionnaire scores | one year
  Effect of patients' age, education, gender, maternal education, nationality on 9-item SDM Questionnaire scores
Effect of treating physicians' age, specialty, years of experience on 9-item SDM Questionnaire scores | one year
  Effect of treating physicians' age, specialty, years of experience on 9-item SDM Questionnaire scores
Effect of patients' Montreal Cognitive Assessment scores on 9-item SDM Questionnaire scores | one year
  Effect of patients' Montreal Cognitive Assessment scores on 9-item SDM Questionnaire scores
Correlation of the 9-item SDM Questionnaire scores with the Client Satisfaction Questionnaire scores | one year
  Correlation of the 9-item SDM Questionnaire scores with the Client Satisfaction Questionnaire scores

CONTACTS AND LOCATIONS:
Overall Officials: Dimitrios Kontis, MD, PHD, Study Director — Psychiatric Hospital of Attica
Locations (1):
- Thriassion General Hospital, Elefsina, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Taking shared decision making more seriously. Lancet. 2011 Mar 5;377(9768):784. doi: 10.1016/S0140-6736(11)60290-0. No abstract available. PMID 21377556
- [Background] Chewning B, Bylund CL, Shah B, Arora NK, Gueguen JA, Makoul G. Patient preferences for shared decisions: a systematic review. Patient Educ Couns. 2012 Jan;86(1):9-18. doi: 10.1016/j.pec.2011.02.004. Epub 2011 Apr 6. PMID 21474265
- [Background] De Las Cuevas C, Penate W, Perestelo-Perez L, Serrano-Aguilar P. Shared decision making in psychiatric practice and the primary care setting is unique, as measured using a 9-item Shared Decision Making Questionnaire (SDM-Q-9). Neuropsychiatr Dis Treat. 2013;9:1045-52. doi: 10.2147/NDT.S49021. Epub 2013 Jul 30. PMID 23950646
- [Background] Flynn KE, Smith MA, Vanness D. A typology of preferences for participation in healthcare decision making. Soc Sci Med. 2006 Sep;63(5):1158-69. doi: 10.1016/j.socscimed.2006.03.030. Epub 2006 May 11. PMID 16697096
- [Background] Kriston L, Scholl I, Holzel L, Simon D, Loh A, Harter M. The 9-item Shared Decision Making Questionnaire (SDM-Q-9). Development and psychometric properties in a primary care sample. Patient Educ Couns. 2010 Jul;80(1):94-9. doi: 10.1016/j.pec.2009.09.034. Epub 2009 Oct 30. PMID 19879711
- [Background] Mah HC, Muthupalaniappen L, Chong WW. Perceived involvement and preferences in shared decision-making among patients with hypertension. Fam Pract. 2016 Jun;33(3):296-301. doi: 10.1093/fampra/cmw012. Epub 2016 Mar 18. PMID 26993483
- [Background] Pollard S, Bansback N, Bryan S. Physician attitudes toward shared decision making: A systematic review. Patient Educ Couns. 2015 Sep;98(9):1046-57. doi: 10.1016/j.pec.2015.05.004. Epub 2015 May 23. PMID 26138158
- [Background] Schneider A, Korner T, Mehring M, Wensing M, Elwyn G, Szecsenyi J. Impact of age, health locus of control and psychological co-morbidity on patients' preferences for shared decision making in general practice. Patient Educ Couns. 2006 May;61(2):292-8. doi: 10.1016/j.pec.2005.04.008. PMID 15896943
- [Background] Smith GL, Volk RJ. Nonclinical Factors Affecting Shared Decision Making. JAMA. 2017 Jul 25;318(4):391. doi: 10.1001/jama.2017.7841. No abstract available. PMID 28742899
- [Background] Stacey D, Legare F, Col NF, Bennett CL, Barry MJ, Eden KB, Holmes-Rovner M, Llewellyn-Thomas H, Lyddiatt A, Thomson R, Trevena L, Wu JH. Decision aids for people facing health treatment or screening decisions. Cochrane Database Syst Rev. 2014 Jan 28;(1):CD001431. doi: 10.1002/14651858.CD001431.pub4. PMID 24470076